CLINICAL TRIAL: NCT03218800
Title: Ertapenem Administered Subcutaneously Versus Intravenously for Urinary Tract Infections in Oncological Palliative Care Patients: a Randomized, Open, Non-inferiority Clinical Trial
Brief Title: Ertapenem Administered Subcutaneously Versus Intravenously
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: not enough participants due to COVID19 pandemia
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Luciana Ramadas, MD, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ertapsubcut
Record Dates: First submitted 2017-07-06; First posted 2017-07-17 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Urinary Tract Infections
Keywords: subcutaneous; ertapenem; urinary tract infection; advanced cancer; palliative care
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Ertapenem (Active Comparator): Patients with urinary tract infection will be treated with ertapenem by the intravenous route.
  Interventions: Combination Product: Ertapenem
- Subcutaneous Ertapenem (Experimental): Patients with urinary tract infection will be treated with ertapenem by the subcutaneous route.
  Interventions: Combination Product: Ertapenem

INTERVENTIONS:
Combination Product: Ertapenem — Dose: 1g per day if creatinine clearance > 30mL/min or 500 mg per day if creatinine clearance < 30mL/min.
  Dilution: 50 ml saline solution. Duration 30 minutes.

SUMMARY:
Infections requiring intravenous antimicrobial therapy are very common events in patients with advanced cancer. Nevertheless, these patients frequently present vascular damages becoming extremely difficult to access and maintain intravenous route for hydration and nutritional support. In this context, the subcutaneous route could be implemented as an alternative route for replacement of fluids, electrolytes and drugs. Few studies have evaluated the possibility of using the subcutaneous route for treatment of infections though.

Patients in palliative care often have infections caused by multidrug resistant bacterial such as beta-lactamase producing bacteria. In this context, we hypothesize Ertapenem subcutaneously is not inferior to the same drug intravenously for the treatment of urinary infections in patients on oncologic palliative care. A non-inferiority clinical trial would be adequate and could provide stronger evidence on the possibility of this alternative route for antibiotic therapy in urinary tract infections, with important advantages such as greater convenience of use.

DETAILED DESCRIPTION:
This is a randomized open label clinical trial to evaluate Ertapenem administered subcutaneously is non-inferior to the same antibiotic intravenously to treat urinary tract infections in oncological palliative care patients.

The study will be performed at the Palliative Care Unit (PCU) of the National Cancer Institute of Brazil José Alencar Gomes da Silva (INCA), a 56-bed hospital and the only public hospital for cancer palliative care located in the city of Rio de Janeiro, Brazil.

A sample of 82 patients was estimated, considering the level of significance (alpha) of unilateral 2.5%, the power of the study (1-beta) of 80%, the non-inferiority limit of 4%, and success percentages in the groups control and experimental studies of 92% and 100%, respectively. Once the high mortality rate of the study site (about 60%, according to unpublished administrative information), it was decided to increase this number by 30% to compensate for possible losses, totaling 106 patients, 53 in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Any type of cancer in palliative care;
* Urinary tract infection;
* Informed consent assigned by the patient or legal representative.

Exclusion Criteria:

* Neutropenia;
* Unconsciousness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
microbiological cure | seven days for cystitis and fourteen days for pyelonephritis
  negative uroculture at the end of the treatment

SECONDARY OUTCOMES:
adverse events | 30 days
  infusion related adverse events
clinical response | 14 days
  improve urinary tract symptoms after ertapenem treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Ramadas, Study Chair — INCA- Instituto Nacional de Câncer
Locations (1):
- INCA Instituto Nacional do Cancer, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forestier E, Gros S, Peynaud D, Levast M, Boisseau D, Ferry-Blanco C, Labe A, Lecomte C, Rogeaux O. [Ertapenem administered intravenously or subcutaneously for urinary tract infections caused by ESBL producing enterobacteriacea]. Med Mal Infect. 2012 Sep;42(9):440-3. doi: 10.1016/j.medmal.2012.07.005. Epub 2012 Aug 25. French. PMID 22925551
- [Background] Frasca D, Marchand S, Petitpas F, Dahyot-Fizelier C, Couet W, Mimoz O. Pharmacokinetics of ertapenem following intravenous and subcutaneous infusions in patients. Antimicrob Agents Chemother. 2010 Feb;54(2):924-6. doi: 10.1128/AAC.00836-09. Epub 2009 Nov 23. PMID 19933804
- [Background] Grigoryan L, Trautner BW, Gupta K. Diagnosis and management of urinary tract infections in the outpatient setting: a review. JAMA. 2014 Oct 22-29;312(16):1677-84. doi: 10.1001/jama.2014.12842. PMID 25335150
- [Background] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Background] Tomera KM, Burdmann EA, Reyna OG, Jiang Q, Wimmer WM, Woods GL, Gesser RM; Protocol 014 Study Group. Ertapenem versus ceftriaxone followed by appropriate oral therapy for treatment of complicated urinary tract infections in adults: results of a prospective, randomized, double-blind multicenter study. Antimicrob Agents Chemother. 2002 Sep;46(9):2895-900. doi: 10.1128/AAC.46.9.2895-2900.2002. PMID 12183244
- See also: ertapenem prescribing information — https://www.merck.com/product/usa/pi_circulars/i/invanz/invanz_pi.pdf
- See also: Power calculator for binary outcome non-inferiority trial — https://www.sealedenvelope.com/power/binary-noninferior/